CLINICAL TRIAL: NCT07380594
Title: Descriptive Study of Psychiatric Symptoms in White-Sutton Syndrome
Acronym: PSY-POGZ
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MOTTOLESE 2025
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: People With White Sutton Syndrome
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with White Sutton syndrome
  Interventions: Other: Interviews; Other: Questionnaires

INTERVENTIONS:
Other: Interviews — An inclusion interview and a second interview 3 to 6 months after the inclusion interview
Other: Questionnaires — K-SADS-PL DSM5 et M.I.N.I 5.0.0 French version / DSM-IV

SUMMARY:
White Sutton syndrome is a rare developmental disorder identified following the description of de novo variations in the POGZ gene, responsible for neurocognitive disorders that may be associated with other signs including hypotonia, deafness, visual disorders, tendency to be overweight, gastrointestinal disorders, convulsions, sleep disorders with sleep apnoea and facial morphological peculiarities. A descriptive study focusing on the neuropsychological assessments of patients showed an absence of systematic intellectual disability and clinical heterogeneity. Psychiatrically, anxiety seems to predominate and manifest itself broadly in the form of generalised anxiety disorder, phobic disorder or obsessive-compulsive disorder. Some patients may also present with autism spectrum disorders, behavioural disorders and attention disorders with or without hyperactivity. Psychiatric symptoms appear to be present in many patients, but with varying frequency and heterogeneous manifestations. Psychiatric manifestations and symptoms can complicate the already complex and often multidisciplinary management of patients. It is therefore essential to define more precisely the psychological characteristics of patients and the psychiatric comorbidities that may be associated with this condition in order to adapt behavioural, environmental and therapeutic management strategies.Psychiatric symptoms appear to be present in many patients, but with varying frequency and heterogeneous manifestations. Psychiatric manifestations and symptoms can complicate the already complex and often multidisciplinary management of patients. It is therefore essential to define more precisely the psychological characteristics of patients and the psychiatric comorbidities that may be associated with this condition in order to adapt behavioural, environmental and therapeutic management strategies. This would make it possible to consider methods for early detection and faster management of psychiatric comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with White Sutton syndrome (genetic mutation identified by genetic testing) adults and children, and French speakers
* Patient or carer able to complete a questionnaire in French lasting 1 to 2 hours
* Age > 6 years (lower age limit for the primary endpoint)
* Consent of the patient (and their parents if the patient is a minor) and legal representative (for patients under guardianship or trusteeship) to participate in the study

Exclusion Criteria:

* Absence of genetic confirmation of the diagnosis
* Refusal by parents or legal representatives to participate or authorise the use of data for research purposes
* Technical impossibility of conducting the interview by videoconference or telephone
* Unfeasible protocol
* patient interruption

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with White Sutton syndrome
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of symptoms and psychiatric diagnoses through a medical interview. | 6 to 9 months
Assessment of symptoms and psychiatric diagnoses through an MINI scales for adults. | 6 to 9 months
Assessment of symptoms and psychiatric diagnoses through a K-SADS scales for children aged 6 to 18. | 6 to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France